CLINICAL TRIAL: NCT03714555
Title: A Phase II Pilot Study of Disulfiram and Copper Gluconate in Patients With Metastatic Pancreatic Cancer and Rising CA-19-9 Levels While Receiving Abraxane-Gemcitabine or FOLFIRINOX or Single-Agent Gemcitabine
Brief Title: Disulfiram-Copper Gluconate in Met Pancreas Cancer w Rising CA19-9 on Abraxane-Gemzar, FOLFIRINOX or Gemcitabine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed due to low subject enrollment at site.
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN-203
Record Dates: First submitted 2018-10-09; First posted 2018-10-22 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Restraint, Physical; 130-nm albumin-bound paclitaxel; Gemcitabine; Clinical Protocols; Disulfiram; Gluconates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nab-Paclitaxel/Gemcitabine + DSF/Cu (Active Comparator): Subjects with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of treatment with Nab-Paclitaxel-Gemcitabine with rising CA 19-9 levels in the absence of radiographic evidence of progression will continue to receive treatment with addition of Disulfiram+Copper Gluconate until disease progression.
  Interventions: Diagnostic Test: Safety Laboratories; Other: AE Assessment; Other: Physical Exam; Other: Concomitant Medication Review; Diagnostic Test: Tumor Imaging; Drug: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate; Drug: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate; Drug: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate
- FOLFIRINOX +DSF/Cu (Active Comparator): Subjects with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of treatment with FOLFIRINOX and with rising CA 19-9 levels in the absence of radiographic evidence of progression will continue to receive treatment with addition of Disulfiram+Copper Gluconate until disease progression.
  Interventions: Diagnostic Test: Safety Laboratories; Other: AE Assessment; Other: Physical Exam; Other: Concomitant Medication Review; Diagnostic Test: Tumor Imaging; Drug: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate; Drug: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate; Drug: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate
- Single-Agent Gemcitabine +DSF/Cu (Active Comparator): Subjects with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of treatment with Single-Agent Gemcitabine and with rising CA 19-9 levels in the absence of radiographic evidence of progression will continue to receive treatment with addition of Disulfiram+Copper Gluconate until disease progression.
  Interventions: Diagnostic Test: Safety Laboratories; Other: AE Assessment; Other: Physical Exam; Other: Concomitant Medication Review; Diagnostic Test: Tumor Imaging; Drug: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate; Drug: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate; Drug: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate

INTERVENTIONS:
Diagnostic Test: Safety Laboratories — Complete blood cell count (CBC) w Differential, comprehensive metabolic panel (CMP), Prothrombin time/international normalized ratio (PT/INR) Activated Partial Thromboplastin Time (aPTT), Urinalysis
Other: AE Assessment — Assessment of Adverse Events (AE)
Other: Physical Exam — Physical Exam, Weight, Vital Signs, Eastern Cooperative Oncology Group (ECOG) Performance Status
Other: Concomitant Medication Review — Prior and Concomitant Medication Review
Diagnostic Test: Tumor Imaging — Tumor CT or MRI
Drug: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate — nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
Drug: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate — FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate dispensing
Drug: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate — Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing

SUMMARY:
This is an open-label Phase 2 Pilot study to evaluate Disulfiram + Copper Gluconate in patients metastatic pancreatic cancer whose CA-19-9 levels rise while receiving nab-paclitaxel (Abraxane) plus gemcitabine (Gemzar) or FOLFIRINOX or single-agent gemcitabine (Gemzar). Patient must have received a minimum of 8 weeks of treatment and have rising CA-19-9 levels in the absence of radiographic evidence of progression.

DETAILED DESCRIPTION:
This study has 3 arms with 5 patients enrolled in each of the three arms. The three treatment arms are based upon whether the patient has previously received Abraxane-Gemcitabine or FOLFIRINOX or single-agent Gemcitabine without radiographic evidence of disease progression for a minimum of 8 weeks , based on the investigator's opinion, but with a rising Carbohydrate antigen 19-9 (CA 19-9) levels. Rising CA 19-9 is defined as an increased over baseline of > 20% in two consecutive time points within 8 days of each other. Study sites will provide all chemotherapy for patients participating in the study as a "standard of care". DSF/Cu (Disulfiram + Copper Gluconate) will be provided by the Sponsor and shipped from the Sponsor's central depot to the study sites. Sufficient amounts of DSF/Cu will be available at the study site prior to enrolling patients in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed adenocarcinoma of the pancreas that is metastatic and for which potential curative measures, such as resection of an isolated metastasis, are not available. Patients with islet cell neoplasms are excluded.
2. Patient should currently be receiving a chemotherapy regimen comprising FOLFIRINOX or Abraxane-Gemcitabine or single-agent Gemcitabine as front-line treatment for metastatic disease. Patients who have had chemotherapy in the adjuvant or neoadjuvant setting are eligible.
3. Patients must have previously received a minimum of 8 weeks of therapy with Abraxane-Gemcitabine or FOLFIRINOX or single-agent Gemcitabine without radiographic evidence of disease progression based on the investigator's opinion, but a rising CA 19-9 level, and still be undergoing treatment with Abraxane-Gemcitabine or FOLFIRINOX or single-agent Gemcitabine. Increased CA 19-9 is defined as an increased over baseline of > 20% in two consecutive time points within 8 days of each other.
4. Patient has one or more metastatic tumors measurable by CT scan. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
5. Male or non-pregnant and non-lactating female and ≥ 18 to ≤ 80 years of age.
6. Patient has adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤ 14 days prior to enrollment) and at Baseline-Day 0: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count ≥ 100,000/mm3 (100 × 109/L); Hemoglobin (Hgb) ≥ 9 g/dL.
7. Patient has the following blood chemistry levels at Screening (obtained ≤ 14 days prior to enrollment) and at Baseline-Day 0:

   * aspartate aminotransferase (AST) (SGOT), Alanine Transaminase (ALT) (SGPT) ≤ 2.5 × upper limit of normal range (ULN), unless liver metastases are present, then ≤ 5 × ULN is allowed. Total bilirubin ≤ 1.5 × ULN.
   * Serum creatinine < 1.5X ULN or estimated creatinine clearance of > 60 mL/min (per Cockroft-Gault formula)
8. Patient has ECOG performance status from 0 to ≤ 1.
9. Patient has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria:

1. Patient has brain metastases.
2. Patient has experienced an increase of ECOG to > 1 between Screening and enrollment.
3. QTc > 480 msec if patient receiving oxaliplatin-containing regimen.
4. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
5. Patient has a history of allergy or hypersensitivity to any of the study drugs, their pharmaceutical class or any of their excipients. The patient exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections of Gemcitabine or Abraxane ® Prescribing Information package inserts or on the Investigator's Brochure for DSF/Cu.
6. Patient has a concomitant serious medical or psychiatric illness that, in the opinion of the investigator, could compromise the patient's safety or the study data integrity.
7. Patient is enrolled in any other clinical protocol or investigational trial involving administration of antineoplastic compounds for the treatment of metastatic pancreatic cancer.
8. Patient is unwilling or unable to comply with study procedures.
9. Abraxane is metabolized by CYP2C8 and CYP3A4. Co-administration of substrates, inhibitors of CYP2C8 (see Appendix C) and/or CYP3A4 (see Appendix D) with Abraxane is not allowed. The following medications and substances are not allowed during the study: ritonavir, saquinavir, indinavir, nelfinavir, rifampicin, carbamazepine, phenytoin, efiravenz, or nerivapine, grapefruit (juice or seeds) or some herbals like St. John's wort.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Jameson, ACNP-BC, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-Paclitaxel/Gemcitabine + DSF/Cu: Subjects with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of treatment with Nab-Paclitaxel-Gemcitabine with rising CA 19-9 levels in the absence of radiographic evidence of progression will continue to receive treatment with addition of Disulfiram+Copper Gluconate until disease progression.
  Safety Laboratories: CBC w Differential, CMP, PT/INR, aPTT, Urinalysis
  AE Assessment: Assessment of Adverse Events
  Physical Exam: Physical Exam, Weight, Vital Signs, ECOG Performance Status
  Concomitant Medication Review: Prior and Concomitant Medication Review
  Tumor Imaging: Tumor CT or MRI
  nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
  FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate dispensing
  Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
- FOLFIRINOX +DSF/Cu: Subjects with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of treatment with FOLFIRINOX and with rising CA 19-9 levels in the absence of radiographic evidence of progression will continue to receive treatment with addition of Disulfiram+Copper Gluconate until disease progression.
  Safety Laboratories: CBC w Differential, CMP, PT/INR, aPTT, Urinalysis
  AE Assessment: Assessment of Adverse Events
  Physical Exam: Physical Exam, Weight, Vital Signs, ECOG Performance Status
  Concomitant Medication Review: Prior and Concomitant Medication Review
  Tumor Imaging: Tumor CT or MRI
  nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
  FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate dispensing
  Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
- Single-Agent Gemcitabine +DSF/Cu: Subjects with metastatic adenocarcinoma of the pancreas who have received a minimum of 8 weeks of treatment with Single-Agent Gemcitabine and with rising CA 19-9 levels in the absence of radiographic evidence of progression will continue to receive treatment with addition of Disulfiram+Copper Gluconate until disease progression.
  Safety Laboratories: CBC w Differential, CMP, PT/INR, aPTT, Urinalysis
  AE Assessment: Assessment of Adverse Events
  Physical Exam: Physical Exam, Weight, Vital Signs, ECOG Performance Status
  Concomitant Medication Review: Prior and Concomitant Medication Review
  Tumor Imaging: Tumor CT or MRI
  nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) Protocol Plus Disulfiram/Copper Gluconate: nab-paclitaxel (Abraxane)/gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
  FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate: FOLFIRINOX regimen Plus Disulfiram/Copper Gluconate dispensing
  Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate: Single-agent gemcitabine (Gemzar) regimen Plus Disulfiram/Copper Gluconate dispensing
Period: Overall Study
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was closed due to low subject enrollment at site.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 1 |  |  | 1
  >=65 years | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  |  | 1
  Male | 0 |  |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 |  |  | 1
  African American | 0 |  |  | 0
  American Indian | 0 |  |  | 0
  Alaska Native | 0 |  |  | 0
  Native Hawaiian | 0 |  |  | 0
  Pacific Rim | 0 |  |  | 0
  Unknown | 0 |  |  | 0
  Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: CA19-9 Plasma Level
Description: Change in plasma CA19-9 level (at least 30%) from baseline
Time Frame: From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Complete Tumor Response
Description: Complete response rate as defined by CT scan using RECIST 1.1 criteria
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Partial Response
Description: Partial response as defined by CT scan using RECIST 1.1 criteria
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Stable Disease
Description: Complete response as defined by CT scan using RECIST 1.1 criteria
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Overall Response Rate
Description: Overall response rate as defined by CT scan using RECIST 1.1 criteria
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Overall Survival
Description: The length of time from the start of treatment that patients are still alive
Time Frame: From date of enrollment until date of death assessed up to 100 months
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Serum Albumin
Description: Change in serum albumin level as a result of treatment
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Body Weight
Description: Change in body weight as a result of treatment
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Muscle Area at the L3 Level - Optional
Description: Change in muscle area at the L3 level using CT scan. Only is L3 is visualized with normally scheduled standard of care CT Scan
Time Frame: as for outcome 1
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Incidence of Toxicities
Description: Physical exam and laboratory testing will be completed and toxicity grading assessed and documented using CTCAE version 4.0
Time Frame: From date of enrollment until the date of follow-up, 30 days after last treatment
Population: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Disulfiram/Copper Gluconate Serum Levels - Area Under the Curve (AUC)
Description: Optional Day 0 (pre-Cycle 1 Day 1) at pre-dose, 2 hours, 4 hours, 24 hours and 4 hours post-dose Cycle 1 Day 7
Time Frame: Day 0 (pre-Cycle 1 Day 1) at pre-dose, 2 hours, 4 hours, 24 hours and 4 hours post-dose Cycle 1 Day 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 Weeks
Description: One patient was treated. This patient was on study for 6 weeks and ended trial participation due to progressive disease.
Arm/Group | Nab-Paclitaxel/Gemcitabine + DSF/Cu | FOLFIRINOX +DSF/Cu | Single-Agent Gemcitabine +DSF/Cu
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel/Gemcitabine + DSF/Cu (N=1) | FOLFIRINOX +DSF/Cu (N=0) | Single-Agent Gemcitabine +DSF/Cu (N=0)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA | NA — Progressive Disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel/Gemcitabine + DSF/Cu (N=1) | FOLFIRINOX +DSF/Cu (N=0) | Single-Agent Gemcitabine +DSF/Cu (N=0)
Transient Flushing/Sweats (Nervous system disorders) | 1 (1) | NA | NA
Muscle Cramp/Burning (Nervous system disorders) | 1 (1) | NA | NA
Depression (Psychiatric disorders) | 1 (1) | NA | NA
Hypertension (Cardiac disorders) | 1 (1) | NA | NA
Headache (Nervous system disorders) | 1 (1) | NA | NA
Slurred Speach (Nervous system disorders) | 1 (1) | NA | NA
Dizziness (Nervous system disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03714555/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT03714555/ICF_001.pdf